CLINICAL TRIAL: NCT03006627
Title: Gender and Opioid Consumption
Acronym: GenderOpioid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GenderOpioids
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Postoperative; Parotitis
MeSH Terms: conditions — Parotitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Male group (Active Comparator): All male patients scheduled for upper abdominal surgeries
  Interventions: Drug: postoperative morphine
- Female group (Active Comparator): All female patients scheduled for upper abdominal surgeries
  Interventions: Drug: postoperative morphine

INTERVENTIONS:
Drug: postoperative morphine — Postoperatively, A loading dose of morphine will be given in incremental doses of 1 mg 5 min apart, till the VAS score reached ≤3. The dose of morphine required to reduce the VAS score to ≤3 will be recorded. Subsequently, PCA pump will be configured to deliver a bolus of 1 mg with a lock-out period lasting for 20 min.

SUMMARY:
Opioids are widely used for pain relief after major abdominal surgeries[1]. Sex differences in the opioid analgesia have been reported and investigated in human subjects and animal models In this study, effects of sex difference on response to opioid analgesics after abdominal surgeries will be assessed regarding; analgesic duration (primary variable), frequency of analgesic requirement, total opioid consumption, Opioid related complications (respiratory depression, Nausea & vomiting, itching, over-sedation, delayed intestinal motility).

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II Cases scheduled for elective intraabdominal surgeries

Exclusion Criteria:

* diabetes,
* postmenopausal females,
* laparoscopic surgery,
* regional anesthesia emergency procedures,
* sepsis,
* hepatectomy,
* Renal impairment, and
* hepatic impairment,
* mental and psychiatric disorders.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
postoperative morphine consumption | 24 hours after surgery

IPD SHARING:
Plan to Share IPD: Undecided